CLINICAL TRIAL: NCT01037894
Title: Can Acupuncture Benefit Surgical Patients With Haemorrhagic Stroke?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GW003
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: Acupuncture,Intracerebral hemorrhage, Stroke
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Acupuncture and conventional rehabilitation
  Interventions: Procedure: Acupuncture
- Control (Active Comparator): Conventional rehabilitation only
  Interventions: Procedure: Conventional rehabilitation

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture from physiotherapist (with accredited training in acupuncture) in Shatin Hospital, three sessions per week for six weeks, and each session 30 minutes.
  Arms: Acupuncture
Procedure: Conventional rehabilitation — In-patient physiotherapy, occupational therapy and speech therapy.
  Arms: Control

SUMMARY:
The purpose is to establish whether acupuncture in addition to conventional rehabilitation programme can improve the functional outcome and quality of life of surgical patients with haemorrhagic stroke, as compared to conventional rehabilitation programme alone.

DETAILED DESCRIPTION:
The investigators aim to recruit 60 patients over a 30 month period. Each patient will have six week of acupuncture treatment (either early within the first six week, or delayed after the first six week of observation and assessment of primary outcome).

Primary outcome measures:

Clinical outcome at the end of week 6 acupuncture treatment: Glasgow Outcome Score extended.

Secondary outcome measures:

Modified Rankin Score, Functional Independence Measure (FIM) score, Modified Aschoff Score, Neurocognitive State Examination (NCSE) score, Barthel index, Modified Rivermead Mobility Index (MRMI), Modified Functional Ambulation Category (MFAC) and motor scores of upper limb and lower limb with Fugl-Meyer Scale at the end of week six acupuncture treatment.

ELIGIBILITY:
Patient inclusion Criteria:

1. Patients after acute hemorrhagic stroke;
2. Within the first month after acute presentation;
3. Premorbid mobility level: Independent Indoor or Outdoor Walker;
4. Co-operative and willing to comply with the rehabilitation program;

Patient exclusion Criteria:

1. Cardiac Pacemaker;
2. Patient who is apprehensive to acupuncture;
3. Clotting abnormality;
4. Poor local skin conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended | Six week

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) score | Six week
Modified Aschoff Score | Six week
Neurocognitive State Examination(NCSE)score | Six week
Motor scores of upper limb and lower limb with Fugl-Meyer Scale | six week
Modified Functional Ambulation Category (MFAC) | Six week
Modified Rivermead Mobility Index (MRMI) | Six week
Barthel Index | Six week
Modified Rankin Scale | Six week

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Division of Neurosurgery, CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China